CLINICAL TRIAL: NCT03819530
Title: A Pilot Study of Micronutrient Supplementation for Child of Urban Poverty Iron Project in Selangor, Malaysia
Brief Title: Child of Urban Poverty Iron Project (CUPIP) - A Pilot Study
Acronym: CUPIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20181056741
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Micronutrient Deficiency; Nutrient Deficiency; Stunting
MeSH Terms: conditions — Anemia, Iron-Deficiency; Growth Disorders | interventions — Vitamins

STUDY DESIGN:
Intervention Model Description: Treatment group: receives baseline deworming medication and daily micronutrient supplementation for 4 months; Control group: receives baseline deworming medication only
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation Group (Experimental): Receives baseline deworming medication. Intervention: receive daily micronutrient supplementation packets- 4 month supply, to be taken every day. Blood iron and anthropometric measurements taken at 0 and 4 months.
  Interventions: Dietary Supplement: Vitamin and Mineral Powder
- Control Group (No Intervention): Receives baseline deworming medication. Blood iron and anthropometric measurements taken at 0 and 4 months.

INTERVENTIONS:
Dietary Supplement: Vitamin and Mineral Powder — Vitamin and mineral nutritional supplement. Each packet is 1g of powder, to be taken with food.
  Other Names: Multiple Micronutrient Powder
  Arms: Supplementation Group

SUMMARY:
The first 1,000 days of life are critical periods for brain development. Proper nutrition lays the foundation for optimal growth, health, and neurodevelopment across the lifespan. Poor nutrition in this vulnerable period has irreversible consequences, including stunting, susceptibility to sickness, reduced school performance and productivity, and impaired intellectual and social development. UNICEF reported in 2018 that among the low cost flat residents in urban areas of the Klang Valley, 15% of children under 5 years old were stunted, 22% underweight, and 23% either overweight or obese.

Will a micronutrient supplementation program improve the growth and iron status of children aged 6 months to 5 years staying in Lembah Subang? Children will be randomized into treatment and control groups. Treatment groups will receive dietary micronutrient supplementation packets. Measurements of height and weight and iron status will be taken at baseline and 4 months later.

DETAILED DESCRIPTION:
This is a pilot study in a single-centre, using a single-blind, two-parallel group, randomized trial conducted amongst children aged 6 months to 5 years residing at PPR Lembah Subang, located in the state of Selangor, Malaysia between October 2019 and February 2020 (4 months). The participants were randomly assigned in a 3:2 treatment-to-control allocation to receive, in addition to the baseline deworming treatment, either daily micronutrient packets for 4 months (intervention arm) or no micronutrient supplementation (control group). This residency area comprises a local population with mixed ethnic makeup and poor socioeconomic status (majority are B40).

We distributed flyers, posters, and leaflets with the help of the community mothers in PPR communities to encourage participation. Registration, informed consent and anthropometric measurements, dietary logs and blood drawn for iron status were taken prior to randomization. All children received a baseline deworming treatment at this point.

The treatment group received baseline deworming medications, a 4-month supply of daily micronutrient supplementation and a compliance monitoring log. The control group only received similar baseline deworming medications without any daily micronutrient supplementation. Only the research investigators and outcome assessors were masked to the treatment status whilst the participants and interventionists research investigators were aware of the assigned intervention.

Primary endpoints assessed in this study are changes in serum ferritin and hemoglobin levels at 0 and 4 months after interventions. The secondary endpoints are changes in age-and-sex standardized height and weight percentile scores at 0 and 4 months after micronutrient supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 years living in PPR Lembah Subang

Exclusion Criteria:

* Ex-premature babies and children with congenital abnormalities resulting in gross impairment
* Children whose caregiver did not consent to participation

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin level between baseline and after 4 months mineral supplementation | First blood test upon enrollment, at 0 months. Second blood test at 4 months
  Blood test for serum ferritin level will be done at enrollment (0 months) and again at end of study period, after 4 months of supplementation (or no supplementation for control group).
Change in reticulocyte hemoglobin level between baseline and after 4 months mineral supplementation | First blood test upon enrollment, at 0 months. Second blood test at 4 months
  Blood test for RET-He level will be done at enrollment (0 months) and again at end of study period, after 4 months of supplementation (or no supplementation for control group).
Change in C-reactive protein level between baseline and after 4 months mineral supplementation | First blood test upon enrollment, at 0 months. Second blood test at 4 months
  Blood test for C-reactive protein level will be done at enrollment (0 months) and again at end of study period, after 4 months of supplementation (or no supplementation for control group).

SECONDARY OUTCOMES:
Change in height (cm) | First height measurement upon enrollment at 0 months. Second height measurement at 6 months.
  Height of child will be measured at baseline (0 months) and after 4 months mineral supplementation (or no supplementation for control group).
Change in weight (kg) | First weight measurement upon enrollment at 0 months. Second weight measurement at 4 months.
  Weight of child will be measured at baseline (0 months) and after 4 months mineral supplementation (or no supplementation for control group).

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Chai See Lum, MD, Principal Investigator — University Malaya, Faculty of Medic
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Not planning to share patient data.

REFERENCES:
- [Derived] Wang CC, Abdul Jalal MI, Song ZL, Teo YP, Tan CA, Heng KV, Low MSY, Anuar Zaini A, Lum LCS. A Randomized Pilot Trial of Micronutrient Supplementation for Under-5 Children in an Urban Low-Cost Flat Community in Malaysia: A Framework for Community-Based Research Integration. Int J Environ Res Public Health. 2022 Oct 25;19(21):13878. doi: 10.3390/ijerph192113878. PMID 36360757